CLINICAL TRIAL: NCT02719067
Title: A Longitudinal Follow-up Imaging Study on Children and Adolescents With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201602058RIN
Record Dates: First submitted 2016-03-10; First posted 2016-03-25 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
Keywords: neuropsychological function; neuroimage; developmental changes
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ASD group: Subjects have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV and ICD-10 criteria
- TD group: Typically developing controls without lifetime ASD or a family history of ASD

SUMMARY:
The significance of this project is the first longitudinal study to investigate the changes of neurocognitive functions of children and adolescents with ASD and to identify the potential neuroimaging endophenotype (biomarkers) for ASD in Asian with advanced imaging technique (Tract-based automatic analysis, TBAA; multi-echo resting-state fMRI in addition to single-echo resting-state fMRI). The success of this project will fill the gap of our understanding of longitudinal changes of brain function by neuropsychological and imaging approaches of ASD in Han Chinese in Taiwan, and is anticipated to facilitate the progress of translational research in ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a common severe, clinically and genetically heterogeneous childhood-onset neurodevelopmental disorder. Due to its high prevalence, typical autistic symptoms, and severe lifelong impairment without effective prevention and treatment, the developmental change of brain functions in individuals with this study has been recognized as one of the key topics of ASD. The goal of this project is to prospectively investigate the stability and changes of brain functions assessed by neuropsychological tests and neuroimages in a cohort of children and adolescents with ASD who had the first assessment 3-5 years ago.

Specific Aims: To investigate the stability and changes of neuropsychological and structural and functional connectivity among children and adolescents with ASD as compared to age- and sex-matched typically developing (TD) controls; and to identify predictors for these neurocognitive changes across a 3-5 follow-up period.

The investigators will prospectively follow up 70 ASDs and 70 TDs for reassessments of clinical symptoms, neuropsychological functions, and structural and functional brain connectivity. The assessments include ASD symptoms (ASD only: Autism Diagnostic Interview-Revised, Autism Diagnostic Observation Scale; all: Social Responsiveness Scale (SRS), Social Communication Questionnaires (SCQ), Autism Spectrum Quotient (AQ)), other psychiatric disorders (The Chinese version of the Kiddie Schedule of Schizophrenia and Affective Disorder Scale-Epidemiologic version, K-SADS-E), neuropsychological functions (Conner's Continuous Performance Test) and MRI assessments (T1 and T2 templates, Diffusion Spectrum Imaging, resting-state fMRI).

ELIGIBILITY:
Inclusion Criteria:

ASD group:

* have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV and ICD-10 criteria, made by board-certificated child psychiatrists and who were clinically diagnosed with ASD confirmed by the ADI-R 3-5 years ago
* ages range from 12 to 20 (i.e., 7-17 years old at the first assessment)
* both parents are Han Chinese
* have complete clinical and behavioral data at the 1st assessment
* participants and their parents consented to participate in this longitudinal study 3-5 years ago for complete assessments at follow-up.

TD group:

* ages range from 12 to 20
* both parents are Han Chinese

Exclusion Criteria:

* comorbidity with DSM-IV-TR or DSM-5 diagnoses of ASD, ADHD, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use
* comorbidity with neurological or systemic disorders
* having a first degree relative who may have ASD based on family history method assessment.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 70 ASDs, aged 12-20, from the cohort of ASD established by previous imaging studies supported by National Science Council(NSC),Taiwan (now Ministry of Science and Technology, MOST), who consented to this follow-up study at their first assessments in 2010-2014 and 70 age-, and sex-matched TD.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Structural neuroimaging | 2 hours
  Using diffusing spectrum imaging (DSI) to assess the structural connectivity in brain circuitries

SECONDARY OUTCOMES:
Neuropsychological functions | 0.5 hour
  Conner's Continuous Performance Test (CCPT) is used to assess the sustained attention, cognitive controls, and vigilance

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan